CLINICAL TRIAL: NCT06522815
Title: Deep Learning Algorithm Update Using Real Patients for Out-of-hospital Obstructive Sleep Apnea Monitoring
Brief Title: Updating Deep Learning Algorithms for OSA Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sky Labs (Industry)
Collaborators: Gangnam Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2022-0207
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea; Obstructive Sleep Apnea-hypopnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Level 1 polysomnography patient (Experimental): For patients undergoing Level 1 polysomnography, simultaneous collection of photoplethysmography (PPG) signals and polysomnography data is performed using the CART-I PLUS device.
  Interventions: Device: CART-I plus; Device: Polysomnography

INTERVENTIONS:
Device: CART-I plus — CART-I PLUS collects signals in two ways:
  ECG: Utilizes the metal on the inner and outer sides as electrodes to detect subtle electrical changes resulting from the contraction and relaxation of the heart muscle.
  PPG: Emits LED light into the blood vessels inside the finger and collects the signal reflected by the blood flow, thereby gathering data on the pulse and functional oxygen saturation (SpO2) of arterial hemoglobin.
  In this clinical trial, PPG signals will be continuously collected during the polysomnography using the PPG method.
Device: Polysomnography — In polysomnography, the following data are collected:
  Electrocardiogram (ECG), Electroencephalogram (EEG), Electromyogram (EMG), Electrooculogram (EOG), Oxygen Saturation (SpO2) Respiratory Analysis, Body Position Monitoring

SUMMARY:
The objective is to enhance the reliability of the algorithm to match that of Level 1 polysomnography by leveraging the diverse data obtained from Level 1 polysomnography to refine the deep learning algorithm.

DETAILED DESCRIPTION:
Patients undergoing Level 1 polysomnography are equipped with the CART-I PLUS device, for collecting polysomnography data alongside concurrent photoplethysmography (PPG) signals.

The collected data is categorized into apnea, hypopnea, and normal segments based on the polysomnography results. Utilizing the PPG and accelerometer (ACC) signals from the CART-I PLUS, metrics such as SaO2 (oxygen saturation), respiratory rate, heart rate (HR), heart rate variability (HRV), and body movement are calculated for each segment. These metrics, along with the PPG and ACC signals, are then used to develop a deep learning model that classifies the segments into apnea, hypopnea, or normal.

Participants are divided into training and validation sets. The deep learning model is trained on data from the participants in the training set, and its performance is evaluated using the validation set.

The algorithm is constructed using convolutional neural networks (CNN), recurrent neural networks (RNN), attention mechanisms, and other advanced techniques recognized for their efficacy in classification tasks, specifically for identifying apnea, hypopnea, and normal segments.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for Level 1 polysomnography at a sleep center who meet all of the following criteria:

* Aged 19 years or older
* Have listened to and understood a thorough explanation of the clinical study and voluntarily agreed to participate

Exclusion Criteria:

* Under 19 years of age
* Unable to collect normal signals during the pre-test or wearing of the CART-I PLUS device
* Refuse to participate in the clinical study
* Have cognitive impairments to the extent that they cannot understand the explanation of the clinical study and therefore cannot make a voluntary decision to participate (e.g., legally incompetent individuals)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-07-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the algorithm and the 95% confidence interval | 11 hours
  Present the accuracy of the algorithm and the 95% confidence interval. If the lower bound of the 95% confidence interval exceeds a minimum accuracy of 0.85, it is considered clinically significant.

SECONDARY OUTCOMES:
Accuracy and 95% confidence intervals for each interval | 11 hours
  Present the accuracy and 95% confidence intervals for each interval. Additionally, precision, recall, ROC curve, and AUC may be presented. The performance comparison between algorithms will use the bootstrap method, and a p-value less than 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Won Joo Kim, MD, PhD, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Arzt M, Young T, Finn L, Skatrud JB, Bradley TD. Association of sleep-disordered breathing and the occurrence of stroke. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1447-51. doi: 10.1164/rccm.200505-702OC. Epub 2005 Sep 1. PMID 16141444
- [Background] Doherty LS, Kiely JL, Swan V, McNicholas WT. Long-term effects of nasal continuous positive airway pressure therapy on cardiovascular outcomes in sleep apnea syndrome. Chest. 2005 Jun;127(6):2076-84. doi: 10.1378/chest.127.6.2076. PMID 15947323
- [Background] Kim J, In K, Kim J, You S, Kang K, Shim J, Lee S, Lee J, Lee S, Park C, Shin C. Prevalence of sleep-disordered breathing in middle-aged Korean men and women. Am J Respir Crit Care Med. 2004 Nov 15;170(10):1108-13. doi: 10.1164/rccm.200404-519OC. Epub 2004 Sep 3. PMID 15347562